CLINICAL TRIAL: NCT02082288
Title: Edessy ICSI Outcome Embryo Score (EIOS) Efficacy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Edessy Mahmoud, al-azhar unversity (assuit), faculty of medicine, obstetrics and gynecology department, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1234
Record Dates: First submitted 2014-03-04; First posted 2014-03-10 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Infertility
Keywords: ICSI outcome
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Edessy ICSI Outcome Embryo Score (Experimental): ICSI
  Interventions: Other: Edessy ICSI Outcome Embryo Score

INTERVENTIONS:
Other: Edessy ICSI Outcome Embryo Score — EIOS:
  Age (ys) >35 (0) 30-35 (1) <30 (2) No of retrived oocyte <5 (0) 5-9 (1) ≥ 10 (2) No of EC embryos <2 (0) 2-4 (1) >4 (2) No of good quality embryos <3 (0) 3-5 (1) >5 (2) No of embryos transferred -------- (0) ≤2 (1) >2 (2)

SUMMARY:
Purpose of this study is to detect outcome of intracytoplasmic sperm injection (ICSI) according to EIOS

DETAILED DESCRIPTION:
A total of 243 infertile couples underwent long GnRH agonist protocol in the ART unit, International Islamic Center for Population Studies and Research (IICPSR), Al-Azhar University.

Embryos which reached the two cell stage at 25-27 hr were classified as EC, and the remaining as Non Early Cleavage embryos (NEC). Embryos were assessed again at 64-68 hours post-ICSI for day three embryo morphology score (Loi et al.,2008). The best two or three embryos, according to day 3 embryo morphology were transferred. Each patient was given a score according to EIOS (female age, number of retrieved oocytes, number of EC embryos, number of good quality embryos and number of embryos transferred).

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 40 years old. BMI >25 - 30 kg/m2. Have two ovaries. Regular cycles. 1st ICSI cycle. Long midluteal GnRH protocol

Exclusion Criteria:

uterine factor as a cause of female factor infertility. pelvic masses or diseases (e.g: endometriosis, fibroids, hydro- salpnix, ...). history of medical disorders (e.g: hypertension, D.M, thyroid dysfunction, liver diseases, renal diseases,...).

azoospermia as a cause of male factor infertility.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 243 (Actual)
Dates: Start 2010-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Edessy, MD, Principal Investigator — Al-Azhar University; Abd-Elnasr M Ali, MD, Principal Investigator — Al-Azhar University; Ahmed Fata, MD, Study Director — Al-Azhar University; Wael M Hamed, MSc, Study Chair — Al-Azhar University
Locations (1):
- International Islamic Center for Population Studies and Research (IICPSR), Al-Azhar university, Cairo, Cairo Governorate, Egypt

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Edessy ICSI Outcome Embryo Score
Started | 243
Completed | 243
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 243 infertile couples, attending the ART unit, International Islamic Center for Population Studies and Research (IICPSR), -Al- Azhar University
Arm/Group | Edessy ICSI Outcome Embryo Score
Number analyzed (Participants) | 243
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.12 (3.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 243
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Pregnancy
Description: A clinical pregnancy will be determined by identifying the presence of a gestational sac at six weeks gestation on transvaginal ultrasonography.
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Edessy ICSI Outcome Embryo Score
Number analyzed (Participants) | 243
participants | 71

ADVERSE EVENTS:
Arm/Group | Edessy ICSI Outcome Embryo Score
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes